CLINICAL TRIAL: NCT05807139
Title: Spironolactone in Alcohol Use Disorder (SAUD): A Double-Blind, Placebo-Controlled, Ascending Dose, Phase 1b Study
Brief Title: Spironolactone in Alcohol Use Disorder (SAUD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 10001546; 001546-DA
Record Dates: First submitted 2023-04-10; First posted 2023-04-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12-11

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Consumption; Alcohol Problems; Alcohol Use Disorder; SPIRONOLACTONE; Mineralocorticoid Receptor
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcohol-Related Disorders | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo 1st visit (Experimental): stage 1: Placebostage 2: 2x50 mg/day spironolactonestage 3: 2x100 mg/day spironolactonestage4: 2x200 mg/day spironolactone
  Interventions: Other: Placebo; Drug: Spironolactone
- Placebo 2nd visit (Experimental): stage 1: 2x50 mg/day spironolactonestage 2: Placebostage3: 2x100 mg/day spironolactonestage 4: 2x200 mg/day spironolactone
  Interventions: Other: Placebo; Drug: Spironolactone
- Placebo 3rd visit (Experimental): stage1: 2x50 mg/day spironolactonestage 2: 2x100 mg/day spironolactonestage 3: Placebostage4: 2x200 mg/day spironolactone
  Interventions: Other: Placebo; Drug: Spironolactone
- Placebo 4th visit (Experimental): Stage1: 2x50 mg/day spironolactoneStage 2: 2x100 mg/day spironolactonestage 3: 2x200 mg/day spironolactonestage 4: Placebo
  Interventions: Other: Placebo; Drug: Spironolactone

INTERVENTIONS:
Other: Placebo — Placebo
Drug: Spironolactone — Spironolactone and its matched placebo will be encapsulated into hard gelatin capsules, in same color, size and taste, to allow blinding.
  Participants will receive 2x50 mg/day, 2x100 mg, and 2x200 mg/day in three sessions (Stages); these Visits always occur in ascending order of dosage. In the remaining session, participants receive the placebo.
  Spironolactone is approved by the FDA, commercially available, and used in clinical practice for the treatment of hypertension, NYHA Class III-IV heart failure, edema in cirrhotic patients, and primary hyperaldosteronism. Comprehensive information about spironolactone, including its pharmacological properties, are provided in the Prescribing Information.

SUMMARY:
Background:

Alcohol use disorder (AUD) affects about 29.5 million people in the United States. Only 3 medicines have been approved by Food and Drug Administration to treat AUD. Researchers want to find better treatments for AUD. Animal studies found that a medicine called spironolactone, may decrease the amount of alcohol the animals drank. Spironolactone is approved to treat high blood pressure, or heart failure in people. It is not approved to treat AUD.

Objective:

To test a medicine (spironolactone) in people who sometimes drink excessive alcohol in order to understand how the body breaks down spironolactone and if there are any side effects in people who drink alcohol while taking this medicine.

Eligibility:

People aged 21 and older with AUD.

Design:

Participants will have 4 separate 7-day stays at a clinic in Baltimore over 2 months. Spironolactone is a capsule you swallow. Participants will take a capsule twice a day for 5 days during each clinic stay. During 1 of their 4 stays, they will take a placebo instead of the medicine. The placebo capsule looks just like the spironolactone capsule but contains no medicine. Participants will not know when they are taking the medicine or the placebo.

Participants will not drink alcohol until day 6 of each clinic stay. Then they will be asked to drink alcohol in a bar-like area in the clinic. Their breath and blood alcohol levels and their well-being will be measured.

Participants will undergo other tests in the clinic:

A DEXA (dual energy X-ray absorptiometry) scan uses X-rays to measure bone density and muscle mass. Participants will lie on an open-top, padded table, then a small arm will scan the full length of their body. The radiation participants will get in this study is about the same as from one regular x-ray.

Blood tests. Participants may feel some discomfort at the site of needle entry.

Electrocardiogram. This test records the heart activity. Sensors are attached to the skin with stickers and removed after a few minutes.

Urine tests. All urine will be collected over a 3-day period during each stay. We will measure the amount of urine, and different hormones and salts in the urine.

Questionnaires and tasks. Participants will answer questions about their alcohol use. They will perform tasks to test mood, craving, mental and physical coordination, and how much they feel an effect from alcohol after drinking.

DETAILED DESCRIPTION:
Study Description:

This study will examine pharmacokinetic (PK) and pharmacodynamic (PD) parameters of spironolactone and alcohol, during concomitant oral administration (0, 100, 200, 400 mg/day spironolactone PO), and test the safety and tolerability of spironolactone, co-administered with alcohol, in individuals with alcohol use disorder (AUD).

Objectives:

Our objective is to assess PK and PD parameters during spironolactone-alcohol co-administration, in individuals with AUD. We will also test the safety, tolerability, and potential drug-alcohol interaction.

Endpoints:

Primary Endpoint:

Spironolactone and alcohol PK during concomitant administration (0, 100, 200, and 400 mg/day spironolactone).

Secondary Endpoints:

1. Assessment of subjective and cognitive effects of acute alcohol administration during concomitant spironolactone treatment (0, 100, 200, and 400 mg/day).
2. Number and severity of adverse events (AEs) experienced, compared between placebo (0 mg/day) and all three spironolactone doses (100, 200, 400 mg/day).
3. PK characteristic of spironolactone active metabolites, canrenone, 7-alpha-thiomethylspirolactone (TMS) and 6beta-hydroxy-7alpha-thiomethylspirolactone (HTMS), before and after administration of alcohol.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to enroll in this study, an individual must meet all of the following criteria:

1. At least 21 years old
2. Alcohol Use Disorder (minimum 2 symptoms on a validated diagnostic tool, e.g., the Mini- International Neuropsychiatric Interview (MINI) or the Structured Clinical Interview for DSM Disorders (SCID))
3. At least four days with >= 4 drinks for females or >= 5 drinks for males during the 28-day period prior to screening, according to alcohol TimeLine Follow Back (TLFB)
4. Most recent Clinical Institute Withdrawal Assessment for Alcohol - revised (CIWA-Ar) score is < 10
5. Able to speak, read, write, and understand English as demonstrated by their ability to understand and sign the consent for the NIDA screening protocol.
6. Female participants must be postmenopausal for at least one year, surgically sterile, or practicing a highly effective method of birth control before entry and throughout the study and must have negative pregnancy tests at each stage. Examples of highly effective methods of birth control include abstinence, hormonal contraceptives (e.g., certain birth control pills, contraceptive patch, vaginal ring, or implants), intrauterine device (IUD), tubal ligation, or vasectomy.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Most recent blood tests: potassium > 5.2 mmol/L; creatinine >= 2 mg/dL; eGFR < 60 mL/min/1.73 m^2, hemoglobin A1c (HbA1c) > 6.5 %
2. Clinically significant and/or symptomatic hyponatremia, hypomagnesemia, hypocalcemia, and hyperuricemia based on Medical Advisory Investigators (MAI) or designee judgment.
3. Known history of clinically significant orthostatic hypotension
4. Known history of hypoaldosteronism, hyperaldosteronism, Addison s disease
5. Diagnosis of NYHA class III-IV heart failure, or unstable cardiovascular conditions (e.g., arrhythmias, clinically significant ECG abnormalities)
6. Current use of any diuretic, angiotensin receptor blocker (ARB), angiotensin converting enzyme inhibitor (ACEI), potassium supplementation, potassium containing salt substitute, heparin and low molecular weight heparin (LMWH), trimethoprim, lithium, digoxin, cholestyramine
7. Current use of MR antagonists
8. Current use of FDA-approved pharmacotherapy for AUD, or seeking treatment for AUD
9. Known history of prior hypersensitivity reaction to spironolactone or other MR antagonists, or any of the product components
10. Known history of alcohol withdrawal seizure and delirium tremens.
11. Physical and/or mental health conditions that are clinically unstable, as determined by the study clinicians, including (but not limited to) major depressive disorder or generalized anxiety disorder unstable during the past three months or other psychiatric conditions (e.g., schizophrenia, bipolar disorder) unstable during the past twelve months prior to screening.
12. Pregnancy, intention to become pregnant, or breastfeeding.
13. Any other reason or clinical condition that the Investigators judge would interfere with study participation and/or be unsafe for a participant.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Describe steady-state PK of spironolactone in individuals with AUD, before and after oral alcohol administration. | Before and after oral alcohol administration.
  PK characteristics of spironolactone (e.g., total concentration, peak concentration, elimination half-life) before (day 5) and after (day 6) oral alcohol administration.
Describe alcohol PK during concomitant spironolactone use | 12 hours after oral alcohol administration
  PK characteristics of alcohol (e.g., blood alcohol concentrations, time for elimination) during concomitant spironolactone treatment (0, 100, 200, and 400 mg/day)

SECONDARY OUTCOMES:
Determine whether spironolactone alters subjective and cognitive effects of acute alcohol administration | 12 hours after oral alcohol administration
  Subjective response to alcohol (e.g., sedation, stimulation, mood) and cognitive performance (e.g., psychomotor function, attention) under alcohol administration, during concomitant spironolactone treatment (0, 100, 200, and 400 mg/day)
Determine safety, tolerability, and potential drug-alcohol interaction by administering spironolactone, combined with alcohol, in individuals with AUD | 12 hours after oral alcohol administration
  Number and intensity of adverse events (AEs) experienced under different spironolactone doses (0, 100, 200, 400 mg/day)
Describe steady-state PK of spironolactone metabolites in individuals with AUD, before and after alcohol administration | Before and after oral administration of alcohol.
  PK characteristics (e.g., total concentration, peak concentration, elimination half-life) of spironolactone metabolites; canrenone, TMS, HTMS, before (day 5) and after (day 6) alcohol administration.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing with other protocols. Data obtained under this protocol and the NIDA screening protocol may be shared and combined for analysis. This will also allow us to avoid repeating assessments that are scheduled in both protocols during the same period of time, therefore avoiding duplication and minimizing participant fatigue. Participants may also consent for other NIH protocols and data collected under those protocols may be combined with data from this protocol for exploratory purposes.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months after publication
Access Criteria: To be determined

REFERENCES:
- [Background] Leko AH, McGinn MA, Farokhnia M. The Mineralocorticoid Receptor: An Emerging Pharmacotherapeutic Target for Alcohol Use Disorder? ACS Chem Neurosci. 2022 Jul 6;13(13):1832-1834. doi: 10.1021/acschemneuro.2c00326. Epub 2022 Jun 24. PMID 35748762
- [Background] Farokhnia M, Rentsch CT, Chuong V, McGinn MA, Elvig SK, Douglass EA, Gonzalez LA, Sanfilippo JE, Marchette RCN, Tunstall BJ, Fiellin DA, Koob GF, Justice AC, Leggio L, Vendruscolo LF. Spironolactone as a potential new pharmacotherapy for alcohol use disorder: convergent evidence from rodent and human studies. Mol Psychiatry. 2022 Nov;27(11):4642-4652. doi: 10.1038/s41380-022-01736-y. Epub 2022 Sep 20. PMID 36123420
- [Background] Palzes VA, Farokhnia M, Kline-Simon AH, Elson J, Sterling S, Leggio L, Weisner C, Chi FW. Effectiveness of spironolactone dispensation in reducing weekly alcohol use: a retrospective high-dimensional propensity score-matched cohort study. Neuropsychopharmacology. 2021 Nov;46(12):2140-2147. doi: 10.1038/s41386-021-01117-z. Epub 2021 Aug 2. PMID 34341493
- [Background] Aoun EG, Jimenez VA, Vendruscolo LF, Walter NAR, Barbier E, Ferrulli A, Haass-Koffler CL, Darakjian P, Lee MR, Addolorato G, Heilig M, Hitzemann R, Koob GF, Grant KA, Leggio L. A relationship between the aldosterone-mineralocorticoid receptor pathway and alcohol drinking: preliminary translational findings across rats, monkeys and humans. Mol Psychiatry. 2018 Jun;23(6):1466-1473. doi: 10.1038/mp.2017.97. Epub 2017 May 2. PMID 28461696
- [Background] Leggio L, Ferrulli A, Cardone S, Miceli A, Kenna GA, Gasbarrini G, Swift RM, Addolorato G. Renin and aldosterone but not the natriuretic peptide correlate with obsessive craving in medium-term abstinent alcohol-dependent patients: a longitudinal study. Alcohol. 2008 Aug;42(5):375-81. doi: 10.1016/j.alcohol.2008.03.128. Epub 2008 May 16. PMID 18486430